CLINICAL TRIAL: NCT01388114
Title: Clinical Evaluation of e- Ab Sensor - Based Real-time Diagnosis of Serum Procalcitonin Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201010020R
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Sepsis
Keywords: Procalcitonin Measurement
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrosensing antibody probing system (e- Ab sensing) (Experimental)
  Interventions: Device: Electrosensing Antibody Probe System (e- Ab sensing)

INTERVENTIONS:
Device: Electrosensing Antibody Probe System (e- Ab sensing) — Electrosensing antibody probing system (e- Ab sensing), which was developed for the rapid and sensitive detection of hapten, proteins or viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti-procalcitonin antibody and procalcitonin in the serum of the patients. The system incorporates the use of engineered semiconductive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe which specifically and selectively binds procalcitonin polypeptide target molecules in the test specimen

SUMMARY:
The purpose of this study is to develop a real-time diagnostic technique with e- Ab sensor for serum PCT level measurement will offer a test with lower cost, and increase the applicability of serum Procalcitonin (PCT) level in daily clinical practice.

DETAILED DESCRIPTION:
Sepsis is a clinical syndrome with complex interactions between microorganism, host immune, inflammatory and coagulation response. The mortality rate associated with septic shock is high, up to 40-70%. Currently, the diagnosis of sepsis depends on microbial infection and systemic inflammatory response syndrome, which lacks sensitivity and specificity. Accordingly, Society of Critical Care Medicine (SCCM) offered new recommendations about the diagnosis of sepsis in 2001, which included the serum level of procalcitonin (PCT). Increased PCT levels through the clinical course correlated with higher mortality in critically-ill patients. On the other hand, recent studies also showed PCT levels could guide the antibiotic treatment in patients with sepsis or lower respiratory tract infection. Besides usage in sepsis population, serum PCT level could also be used for aids in diagnosis of bacterial infection and for guide of antibiotic treatment in acute exacerbation of chronic obstructive airway disease. However, current method of PCT assay depends on the Kryptor system developed by BRAHMS, Germany, with the functional sensitivity of 60 pg/mL. Each assay costs 1300 NT dollars, which is too expensive for serial follow-up of serum PCT levels. A real-time diagnostic technique with e- Ab sensor for serum PCT level measurement will offer a test with lower cost, and increase the applicability of serum PCT level in daily clinical practice. Here, the investigators conduct a study to develop a real-time diagnostic technique with e- Ab sensor for serum PCT level measurement in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to medical intensive care units

Exclusion Criteria:

* Patients who refuse consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Performance of e- Ab sensor for serum PCT level measurement | 1 Day
  The serum procalcitonin level from e- Ab sensor would be compared with the results from Kryptor assay system, Brahms, Germany. The correlation between serum procalcitonin levels from e- Ab sensor and from Kryptor assay system would be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, MD, PhD, Principal Investigator — National Taiwan Universtiy Hospital
Locations (1):
- National Taiwan University Hosital, Taipei, Taiwan